CLINICAL TRIAL: NCT05162586
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging, Parallel and Adaptive Study to Evaluate the Efficacy and Safety of Enpatoran in SLE and in CLE (SCLE and/or DLE) Participants Receiving Standard of Care (WILLOW)
Brief Title: The WILLOW Study With M5049 in SLE and CLE (SCLE and/or DLE) (WILLOW)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200569_0003; 2021-004648-27 (EudraCT Number); 2024-510872-18-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-08; First posted 2021-12-17 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Toll-like Receptor 7; Toll-like Receptor 8; WILLOW; Adults; SLE; CLE; Lupus; Discoid lupus erythematosus; Subacute cutaneous lupus erythematosus; M5049; Enpatoran
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A: Placebo (Placebo Comparator): Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (Cutaneous Lupus Erythematosus Disease Area and Severity Index [CLASI-A] greater than or equal to [>=] 8) will be enrolled in Cohort A to receive placebo matched to Enpatoran.
  Interventions: Drug: Placebo
- Cohort A: Enpatoran low dose (Experimental): Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (CLASI-A >= 8) will be enrolled in Cohort A to receive low dose of Enpatoran.
  Interventions: Drug: Enpatoran low dose
- Cohort A: Enpatoran medium dose (Experimental): Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (CLASI-A >= 8) will be enrolled in Cohort A to receive medium dose of Enpatoran.
  Interventions: Drug: Enpatoran medium dose
- Cohort A: Enpatoran high dose (Experimental): Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (CLASI-A >= 8) will be enrolled in Cohort A to receive high dose of Enpatoran.
  Interventions: Drug: Enpatoran high dose
- Cohort B (Part 1 + Part 2): Placebo (Placebo Comparator): Participants with active SLE who have moderate to high systemic disease activity (British Isles Lupus Assessment Group [BILAG A/2B]) with 1 or 2 of the following: CLASI-A >= 8 and/or Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) >= 6 will be enrolled in Cohort B to receive placebo matched to Enpatoran .
  Interventions: Drug: Placebo
- Cohort B (Part 1 + Part 2): Enpatoran high dose (Experimental): Participants with active SLE who have moderate to high systemic disease activity (BILAG A/2B) with 1 or 2 of the following: CLASI-A >= 8 and/or SLEDAI >= 6 will be enrolled in Cohort B to receive high dose of Enpatoran.
  Interventions: Drug: Enpatoran high dose
- Cohort B (Part 2): Enpatoran low dose (Experimental): Participants with active SLE who have moderate to high systemic disease activity (BILAG A/2B) with 1 or 2 of the following: CLASI-A >= 8 and/or SLEDAI >= 6 will be enrolled in Cohort B to receive low dose of M5049.
  Interventions: Drug: Enpatoran low dose
- Cohort B (Part 2): Enpatoran medium dose (Experimental): Participants with active SLE who have moderate to high systemic disease activity (BILAG A/2B) with 1 or 2 of the following: CLASI-A >= 8 and/or SLEDAI >= 6 will be enrolled in Cohort B to receive medium dose of Enpatoran.
  Interventions: Drug: Enpatoran medium dose

INTERVENTIONS:
Drug: Enpatoran low dose — Participants will receive film-coated tablets of Enpatoran at a low dose orally, twice daily (BID) up to 24 weeks.
  Other Names: M5049
  Arms: Cohort A: Enpatoran low dose; Cohort B (Part 2): Enpatoran low dose
Drug: Enpatoran medium dose — Participants will receive film-coated tablets of Enpatoran at a medium dose, orally, BID up to 24 weeks.
  Other Names: M5049
  Arms: Cohort A: Enpatoran medium dose; Cohort B (Part 2): Enpatoran medium dose
Drug: Enpatoran high dose — Participants will receive film-coated tablets of Enpatoran at a high dose, orally, BID up to 24 weeks.
  Other Names: M5049
  Arms: Cohort A: Enpatoran high dose; Cohort B (Part 1 + Part 2): Enpatoran high dose
Drug: Placebo — Participants will receive placebo matched to Enpatoran up to 24 weeks.
  Arms: Cohort A: Placebo; Cohort B (Part 1 + Part 2): Placebo

SUMMARY:
The purpose of this Proof of Concept (PoC) and Dose-finding (DF) basket study is to evaluate the efficacy and safety of orally administered Enpatoran over 24 weeks in systemic lupus erythematosus (SLE) and cutaneous lupus erythematosus (CLE; subacute cutaneous lupus erythematosus [SCLE] and/or discoid lupus erythematosus [DLE]) participants in a randomized, double-blind, placebo-controlled, parallel, adaptive and dose-ranging setting. Study Duration: 33 weeks Visit Frequency: every 2 or 4 weeks Enpatoran is not available through an expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Active CLE (SCLE and/or DLE) with a CLE disease area and activity index (CLASI-A) >= 8
* Active SLE with presence of: CLASI-A >= 8 and BILAG 2004 1B, C, D (that is [i.e.], No BILAG 2004 A and No BILAG 2004 >= 2B) or BILAG 2004 >= 1A or 2B and 1 or 2 of the following: Hybrid Safety of Estrogens in Systemic Lupus Erythematosus National Assessment (SELENA)-SLEDAI >= 6 at Screening Visit and confirmed clinical hybrid SELENA-SLEDAI >= 4 (excluding laboratory parameters) at Day 1 Visit and/or CLASI-A >= 8
* Receiving a stable dose of at least one of the following standards of care therapies for lupus: Immunomodulator/immunosuppressant, oral corticosteroids, and/or topical corticosteroids
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Autoimmune or rheumatic disease other than SLE or CLE
* Dermatological diseases other than cutaneous manifestations of SLE or CLE
* Uncontrolled medical conditions including significant cardiovascular events, active lupus nephritis, and active neurological disorder
* Ongoing or active clinically significant viral, bacterial, or fungal infection
* History of uncontrolled seizures or other neurological disorder
* History of or positive for human immunodeficiency virus, hepatitis C virus, or hepatitis B virus
* History of malignancy
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (153):
- United States (14):
  - The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Advance Medical Research Center, Miami, Florida
  - New Horizon Research Center, Inc, Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - HMD Research, LLC, Orlando, Florida
  - D&H Tamarac Research Center, LLC, Tamarac, Florida
  - RNA America Health Sciences, Sugar Hill, Georgia
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - AA MRC LLC Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Across the Life Span, Smithfield, North Carolina
  - Ohio State University - CTMO Parent, Columbus, Ohio
  - Ramesh C Gupta, MD - Memphis, TN, Memphis, Tennessee
- Argentina (12):
  - CINME - Centro De Investigaciones Metabolicas, Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Centro Dermatologico Schejtman, Ciudad Autonoma Buenos Aires
  - Hospital Militar Central Dr. Cosme Argerich, Ciudad Autonoma Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata - CIM, Mar del Plata
  - Instituto de Reumatologia, Mendoza
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Instituto Medico de alta Complejidad San Isidro S.A (IMAC), San Fernando
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
  - PSORIAHUE-Medicina Interdisciplinar, San Miguel
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
- Australia (3):
  - Monash Medical Centre Clayton, Clayton
  - Westmead Hospital - SUPERSEDED, Westmead
  - Veracity Clinical Research, Woolloongabba
- Brazil (11):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Oncovida - Centro de Onco-Hematologia de Mato Grosso, Cuiabá
  - CETI - Centro de Estudos em Terapias Inovadoras Ltda., Curitiba
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora
  - Hospital Bruno Born, Lajeado
  - Hospital Moinhos de Vento, Porto Alegre
  - Clínica SER da Bahia, Salvador
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto - CIP - Centro Integrado de Pesquisa, São José do Rio Preto
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo
- Bulgaria (6):
  - DCC 'Sveti Georgi' EOOD - Cardiology Office, Haskovo
  - MC Artmed OOD, Plovdiv
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - DCC "Alexandrovska", EOOD, Sofia
  - Military Medical Academy - MHAT - Sofia - Department of Rheumatology, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD - Clinic of Rheumatology, Sofia
- Chile (6):
  - Clínica Alemana de Osorno, Osorno
  - BioMedica Research Group - Psicomedica Clinical and Research Group, Santiago
  - CeCim Biocinetic, Santiago
  - Centro Medico Prosalud, Santiago
  - CIEC - Centro Internacional de Estudios Clínicos - Valenzuela Y Compania Ltda, Santiago
  - Dermacross, Santiago
- China (20):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Peking Union Medical College Hospital - Beijing Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The 2nd Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital - Oncology, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Hospital for Skin Diseases, Chinese Academy of Medical Sciences, Nanjing
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing
  - Huashan Hospital, Fudan University, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Skin Disease Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- Colombia (5):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas CIREEM S.A.S., Bogotá
  - Servimed S.A.S., Bucaramanga
  - Centro Integral de Reumatologia del Caribe SAS CIRCARIBE SAS, Medellín
  - Healthy Medical Center, Zipaquirá
- Greece (6):
  - "Andreas Syggros" Hospital - Department of Dermatology, Athens
  - General Hospital of Athens Laiko, Athens
  - University Hospital of Patra, Pátrai
  - General Hospital of Thessaloniki "Hippokration", Thessaloniki
  - General Hospital Papageorgiou, Thessaloniki
  - Skin and Venereal Diseases' Hospital, Thessaloniki
- Chaim Sheba Medical Center - pt, Ramat Gan, Israel
- Japan (12):
  - NHO Asahikawa Medical Center - Dept of Gastroenterology, Asahikawa-shi
  - NHO Chibahigashi National Hospital - Dept of Allergy/Rheumatology, Chiba
  - St. Luke's International Hospital - Dept of Immunology/Allergy, Chūōku
  - Hiroshima University Hospital - Dept of Rheumatology/Immunology, Hiroshima
  - Eiraku Clinic - Dept of Rheumatology, Kagoshima
  - Kanazawa University Hospital - Dept of Rheumatology/Immunology, Kanazawa
  - Saitama Medical Center - Dept of Rheumatology/Immunology, Kawagoe-shi
  - Kagawa University Hospital - Dept of Immunology/ Rheumatology, Kita-gun
  - Toho University Ohashi Medical Center - Dept of Immunology/Rheumatology, Meguro-ku
  - Hokkaido University Hospital - Dept of Internal Medicine 2(Rheumatology/Immunolog, Sapporo
  - Tohoku University Hospital - Dept of Hematology/Immunology, Sendai
  - Ehime University Hospital - Dept of Immunology/Rheumatology, Toon-shi
- CAP Research Ltd, Quatre Bornes, Mauritius
- Mexico (11):
  - Consultorio Particular del Dr. Miguel Cortes Hernandez - (dentro del Centro de Especialidades Medicas Vista, Cuernavaca
  - Centro de Estudios de Investigacion Basica y Clinica SC, Guadalajara
  - Centro Medico del Angel, Mexicali
  - CAIMED Investigacion en salud S.A de C.V., Mexico City
  - Centro de Investigacion Clínica GRAMEL S.C, México
  - Citer, Centro de Investigación Y Tratamiento de Las Enfermedades Reumaticas Sa de Cv, México
  - Clinstile, S.A. de C.V., México
  - Consultorio de Reumatologia - Hospital Angeles Lindavista Cons. 445B, México
  - Grupo Medico Camino S.C., México
  - CIMAB S.A. de C.V. - Centro de Investigacion Medica Alberto Bazzoni, Torreón
  - Medical Care & Research SA de CV, Yucatán
- ICS ARENSIA Exploratory Medicine SRL - Republican Clinical Hospital "Timofei Mosneaga", Chisinau, Moldova
- Philippines (7):
  - Perpetual Succour Hospital, Cebu City
  - Davao Doctors Hospital - Medicine, Davao City
  - Iloilo Doctors Hospital, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Chinese General Hospital & Medical Center, Manila
  - Far Eastern University - Dr. Nicanor Reyes Medical Foundation - Department of Child Health, Quezon City
  - Ospital Ng Makati, Quezon City
- Poland (8):
  - Nova Reuma Spolka Partnerska, Bialystok
  - Prywatna Praktyka Lekarska prof Pawel Hrycaj, Kościan
  - Centrum Medyczne Plejady, Krakow
  - Centrum Nowoczesnych Terapii Dobry Lekarz, Krakow
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - Twoja Przychodnia PCM, Poznan
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Clinical Best Solutions - Warszawa, Warsaw
- Romania (6):
  - Centrul Medical Monza SRL - Arensia Exploratory Medicine, Bucharest
  - S.C Delta Health Care S.R.L - Ponderas Academic Hospital, Bucharest
  - Spitalul Clinic "Sf. Maria" - Clinica de Medicina Interna si Reumatologie, Bucharest
  - Spitalul Clinic "Sf. Maria" - parent, Bucharest
  - Spitalul Clinic Colentina - parent, Bucharest
  - Sc Medaudio-Optica SRL, Râmnicu Vâlcea
- Serbia (5):
  - Institute of Rheumatology- 1, Belgrade
  - Institute of Rheumatology-1, Belgrade
  - Institute of Rheumatology, Belgrade
  - University Clinical Center of Serbia - Clinic of Alergology and Imunology, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- South Africa (3):
  - Arthritis Clinical Research Trial Unit - Dr CE Spargo and Dr RB Bhorat, Cape Town
  - University of Pretoria Clinical Research Unit - Parent, Pretoria
  - Naidoo, A - Netcare Umhlanga Hospital, Umhlanga
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña - Servicio de Reumatologia, A Coruña
  - Hospital General de Castellon - Servicio de Reumatologia, Castelló
  - Hospital Universitario 12 de Octubre - Servicio de Reumatologia, Madrid
  - Hospital Regional Universitario de Malaga - Reumatology Dept, Málaga
  - Hospital Universitario Marques de Valdecilla - Servicio de Reumatologia, Santander
  - Hospital Quironsalud Sagrado Corazon - Reumatologia, Seville
  - Hospital Universitario Dr. Peset - Servicio de Reumatologia, Valencia
  - Hospital Universitario Rio Hortega - Servicio de Medicina Interna, Valladolid
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Cheng Hsin General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0003
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Placebo: Participants with cutaneous lupus erythematosus (CLE) (active subacute cutaneous lupus erythematosus [SCLE] and/or discoid lupus erythematosus [DLE]) or systemic lupus erythematosus (SLE) with predominantly active lupus rash (Cutaneous Lupus Erythematosus Disease Area and Severity Index [CLASI-A] greater than or equal to [>=] 8) were enrolled in Cohort A to receive placebo matched to Enpatoran twice daily for 24 weeks.
- Cohort A: Enpatoran 25 mg: Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (CLASI-A >= 8) were enrolled in Cohort A to receive 25 milligrams (mg) of Enpatoran twice daily for 24 weeks.
- Cohort A: Enpatoran 50 mg: Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (CLASI-A >= 8) were enrolled in Cohort A to receive 50 mg of Enpatoran twice daily for 24 weeks.
- Cohort A: Enpatoran 100 mg: Participants with CLE (active SCLE and/or DLE) or SLE with predominantly active lupus rash (CLASI-A >= 8) were enrolled in Cohort A to receive 100 mg of Enpatoran twice daily for 24 weeks.
- Cohort B (Part 1 + Part 2): Placebo: Participants with active SLE who have moderate to high systemic disease activity (British Isles Lupus Assessment Group [BILAG A/2B]) with 1 or 2 of the following: CLASI-A >= 8 and/or Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) >= 6 were enrolled in Cohort B to receive placebo matched to Enpatoran twice daily for 24 weeks during Part 1 and Part 2.
- Cohort B (Part 2): Enpatoran 25 mg: Participants with active SLE who have moderate to high systemic disease activity (BILAG A/2B) with 1 or 2 of the following: CLASI-A >= 8 and/or SLEDAI >= 6 were enrolled in Cohort B to receive 25 mg of Enpatoran twice daily for 24 weeks.
- Cohort B (Part 2): Enpatoran 50 mg: Participants with active SLE who have moderate to high systemic disease activity (BILAG A/2B) with 1 or 2 of the following: CLASI-A >= 8 and/or SLEDAI >= 6 were enrolled in Cohort B to receive 50 mg of Enpatoran twice daily for 24 weeks.
- Cohort B (Part 1 + Part 2): Enpatoran 100 mg: Participants with active SLE who have moderate to high systemic disease activity (BILAG A/2B) with 1 or 2 of the following: CLASI-A >= 8 and/or SLEDAI >= 6 were enrolled in Cohort B to receive 100mg of Enpatoran twice daily for 24 weeks during Part 1 and Part 2.
Period: Overall Study
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Started | 26 | 24 | 26 | 26 | 95 | 71 | 74 | 114
Participants With BILAG≥1A/2B Randomized in Error Due to Systemic Disease Activity | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Cohort B Part 1 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 40
Cohort B Part 2 | 0 | 0 | 0 | 0 | 74 | 71 | 74 | 74
Completed | 22 | 23 | 25 | 24 | 79 | 64 | 65 | 104
Not Completed | 4 | 1 | 1 | 2 | 16 | 7 | 9 | 10
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Not completed — Non-Compliance | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 7 | 6 | 2 | 2
Not completed — Adverse Event | 2 | 0 | 1 | 2 | 4 | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants randomized in the cohort to which they were eligible. Participants who were randomized in error were excluded from FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg | Total
Number analyzed (Participants) | 26 | 23 | 25 | 26 | 94 | 71 | 74 | 114 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11.0) | 42 (12.1) | 47 (14.6) | 45 (14.3) | 42 (12.3) | 42 (12.4) | 39 (12.3) | 44 (12.2) | 42 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 19 | 19 | 87 | 69 | 69 | 110 | 412
  Male | 4 | 6 | 6 | 7 | 7 | 2 | 5 | 4 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 11 | 11 | 47 | 37 | 37 | 51 | 213
  Not Hispanic or Latino | 16 | 14 | 14 | 15 | 47 | 34 | 37 | 63 | 240
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 2 | 3 | 27 | 22 | 18 | 28 | 107
  Asian | 7 | 8 | 9 | 8 | 26 | 16 | 20 | 27 | 121
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 2 | 1 | 3 | 6 | 6 | 3 | 26
  White | 11 | 11 | 12 | 14 | 35 | 24 | 29 | 51 | 187
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index-A (CLASI-A) Total Score at Week 16
Description: The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index) was a validated instrument used to assess disease activity (CLASI-A) and damage in lupus erythematosus. The activity scale included erythema, scale/hypertrophy, active alopecia, recent hair loss, and mucous membrane disease, while the damage scale measured dyspigmentation, atrophy, and scarring. CLASI-A scores ranged from 0 to 70, with mild, moderate, and severe disease corresponding to scores of 0-9, 10-20, and 21-70, respectively. Erythema and scale/hypertrophy sub-scores were computed across 13 body areas, with maximum scores of 39 and 26, respectively. The remaining 5 points reflected contributions from active alopecia (0-3), recent hair loss (0-1), and mucous membrane involvement (0-1), completing the total CLASI-A activity score. Directionality reflected worsening with higher scores and improvement with lower scores.
Time Frame: Baseline, week 16
Population: The Full Analysis Set (FAS) included all participants randomized in the cohort to which they were eligible. Participants who were randomized in error were excluded from FAS. "Overall number of participants analyzed" refers to those evaluable for the outcome measure,
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg
Number analyzed (Participants) | 23 | 22 | 24 | 25
scores on a scale | -5.0 (3.94) | -9.0 (4.60) | -10.2 (6.77) | -9.7 (5.84)

2. Primary Outcome: Cohort B: Number of Participants With British Isles Lupus Assessment Group (BILAG)-Based Composite Lupus Assessment (BICLA) Response at Week 24
Description: BILAG-based BICLA response is defined as participants meeting all of the following criteria: 1. Improvement in baseline BILAG scores in all organ systems with moderate or severe disease activity-i.e., all grade A scores (severe disease requiring high-dose therapy) must improve to B (moderate), C (mild), or D (no activity); all grade B scores (moderate disease requiring moderate therapy) must improve to C or D; 2. No new BILAG A scores and no more than one new BILAG B score; 3. No worsening in total SLEDAI-2K score from baseline; 4. No significant deterioration (≤10%) in physician's global assessment; and 5. No treatment failure, defined as initiation of non-protocol therapy. Directionality is toward clinical improvement and disease stabilization.
Time Frame: At Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 95 | 71 | 74 | 114
Participants | 37 | 41 | 36 | 56

3. Secondary Outcome: Cohort A and B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events (AEs) of Special Interest
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether considered related to the medicinal product or protocol-specified procedure. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAE was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious TEAEs and non-serious TEAEs. Adverse events of special interest (AESI) are serious or non-serious AEs that are of clinical interest and were closely followed.
Time Frame: From screening upto safety follow up period (up to approximately 33 weeks)
Population: The Safety Analysis Set (SAF) included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 26 | 24 | 26 | 26 | 95 | 71 | 74 | 114
Participants
  TEAEs | 12 | 15 | 15 | 21 | 61 | 42 | 47 | 70
  Serious TEAEs | 1 | 2 | 0 | 1 | 3 | 1 | 3 | 5
  AESI | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 3

4. Secondary Outcome: Cohort A and B: Number of Participants With Abnormal Laboratory Parameters
Description: Laboratory parameters included hematology, biochemistry, Urinalysis, Renal Toxicity and Hepatotoxicity. Number of Participants with Abnormal laboratory parameters (severity of grade greater or equal to 3) were reported. Severity of grade 3 or higher TEAEs were graded using National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 toxicity grades, as follows: Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: From screening upto safety follow up period (up to approximately 33 weeks)
Population: The Safety Analysis Set (SAF) included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 26 | 24 | 26 | 26 | 95 | 71 | 74 | 114
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Cohort A and B: Number of Participants With Clinically Important Increases in QT Interval Corrected Using Fridericia's Formula (QTcF)
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, and QT interval. The corrected QT interval (QTcF) was calculated using Fridericia's formula. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semisupine position. Clinical importance was determined by the investigator. The number of participants with clinically important increases in QTCF findings were reported.
Time Frame: From screening upto safety follow up period (up to approximately 33 weeks)
Population: The Safety Analysis Set (SAF) included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 26 | 24 | 26 | 26 | 95 | 71 | 74 | 114
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Cohort A and Cohort B: Change From Baseline in Cutaneous Lupus Activity Investigator's Global Assessment (CLA-IGA) Scale Score at Week 16 and Week 24
Description: The Cutaneous Lupus Activity Investigator's Global Assessment (CLA-IGA) is a validated clinician-reported outcome measure used to assess disease severity in participants with cutaneous lupus erythematosus. It is based on a 5-point ordinal scale that evaluates overall lesion characteristics, where 0 indicates "clear" skin and 4 represents "severe" disease. The scale includes the following categories: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), and 4 (severe).
Time Frame: Baseline and at Week 16 and Week 24
Population: The FAS included all participants randomized in the cohort to which they were eligible. "Overall number of participants analyzed" refers to those evaluable for the outcome measure, while "number analyzed" refers to those evaluable at specific timepoints. Participants who were randomized in error were excluded from FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 26 | 23 | 25 | 26 | 41 | 29 | 38 | 54
units on a scale
  Baseline | 3.0 (0.66) | 3.0 (0.714) | 3.0 (0.61) | 3.179 (0.59) | 2.8 (0.72) | 2.9 (0.67) | 2.7 (0.65) | 2.8 (0.57)
  Week 16: number analyzed (Participants) | 23 | 22 | 24 | 25 | 36 | 27 | 35 | 49
  Week 16 | -0.9 (1.01) | -1.7 (1.09) | -1.5 (1.14) | -1.8 (0.88) | -0.6 (0.96) | -1.1 (1.15) | -1.2 (1.01) | -1.5 (1.00)
  Week 24: number analyzed (Participants) | 20 | 22 | 23 | 24 | 36 | 25 | 36 | 52
  Week 24 | -0.9 (1.17) | -1.8 (0.92) | -1.7 (0.92) | -2.1 (1.08) | -0.8 (1.00) | -1.5 (1.19) | -1.4 (0.94) | -1.8 (0.98)

7. Secondary Outcome: Cohort A and Cohort B: Change From Baseline in Physician's Global Assessment of Cutaneous Lupus Disease Activity Score at Week 16 and 24
Description: The Physician's Global Assessment of Disease Activity was recorded using the 100 millimeter horizontal Visual Analog Scale (VAS). The score reflects the clinician's integrated judgment based on clinical signs, symptoms, laboratory findings, and patient-reported outcomes. PGA is used to quantify disease severity and monitor treatment response over time. Physician rated participant's disease activity on a scale ranged from 0-100 millimeter (mm), where 0 indicated no disease activity and 100 represented maximum disease activity.
Time Frame: Baseline and at Week 16 and Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 26 | 23 | 25 | 25 | 39 | 28 | 35 | 50
millimeter
  Baseline | 61.4 (14.08) | 61.8 (15.37) | 56.3 (19.42) | 61.7 (18.04) | 55.7 (17.08) | 56.1 (15.65) | 56.7 (14.85) | 57.4 (17.42)
  Week 16: number analyzed (Participants) | 23 | 22 | 23 | 24 | 35 | 26 | 32 | 44
  Week 16 | -25.3 (20.55) | -42.5 (23.67) | -35.2 (25.70) | -42.0 (22.94) | -16.7 (20.01) | -26.1 (17.62) | -30.7 (22.78) | -36.0 (22.08)
  Week 24: number analyzed (Participants) | 20 | 22 | 23 | 23 | 35 | 24 | 33 | 48
  Week 24 | -23.9 (25.45) | -44.0 (21.97) | -41.2 (25.12) | -49.1 (22.44) | -21.3 (18.35) | -33.0 (19.68) | -34.8 (20.06) | -39.1 (23.16)

8. Secondary Outcome: Cohort B: Number of Participants With Both BICLA Response and With Clinically Meaningful Corticosteroids (CS) Reduction
Description: BICLA (BILAG-Based Composite Lupus Assessment) defines response as improvement in all baseline BILAG A scores to B, C, or D and all B scores to C or D, with no new A scores and no more than one new B score. Responders must also show no worsening in SLEDAI-2K or Physician's Global Assessment (defined as ≥0.3-point increase). Corticosteroid (CS) reduction is defined as a decrease in daily prednisone-equivalent dose from ≥10 mg at Day 1 to ≤5 mg by Week 12, sustained through Week 24. BILAG grades reflect disease severity: A = severe disease requiring high-dose therapy; B = moderate disease requiring moderate therapy; C = mild stable disease; D = no current activity.
Time Frame: At week 24 (BICLA Response) and Day 1 upto Week 24 (CS Reductions)
Population: The FAS included all participants randomized in the cohort to which they were eligible. "Overall number of participants analyzed" refers to those evaluable for the outcome measure. Participants who were randomized in error were excluded from FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 51 | 34 | 36 | 59
Participants | 16 | 20 | 20 | 28

9. Secondary Outcome: Cohort A and B: Number of Participants With Clinically Meaningful Corticosteroids (CS) Reduction
Description: CS reduction is defined as the reduction of daily prednisone-equivalent dose from >= 10 mg at Day 1 to <= 5 mg by the Week 12 visit and sustained through Week 24. The number of participants with Clinically Meaningful CS Reduction were reported.
Time Frame: Day 1 up to Week 24
Population: The FAS included all participants randomized in the cohort to which they were eligible. Participants who were randomized in error were excluded from FAS. "Overall number of participants analyzed" refers to those evaluable for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 26 | 23 | 25 | 26 | 51 | 34 | 36 | 59
Participants | 6 | 7 | 12 | 9 | 36 | 28 | 27 | 41

10. Secondary Outcome: Cohort A: Number of Participants With CLA-IGA Score 0 or 1 at Week 16 and Week 24
Description: The Cutaneous Lupus Activity Investigator's Global Assessment (CLA-IGA) is a validated clinician-reported outcome measure used to assess disease severity in participants with cutaneous lupus erythematosus. It is based on a 5-point ordinal scale that evaluates overall lesion characteristics, where 0 indicates "clear" skin and 4 represents "severe" disease. The scale includes the following categories: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), and 4 (severe). The number of participants with CLA-IGA score 0 or 1 at Week 16 and Week 24 were reported.
Time Frame: At Week 16 and Week 24
Population: The FAS included all participants randomized in the cohort to which they were eligible. Participants who were randomized in error were excluded from FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg
Number analyzed (Participants) | 26 | 23 | 25 | 26
Participants
  Week 16 | 4 | 10 | 10 | 12
  Week 24 | 7 | 11 | 12 | 14

11. Secondary Outcome: Cohort B: Number of Participants With Systemic Lupus Erythematosus Responder Index-4 (SRI-4) Response at Week 24
Description: SRI-4 response was defined as >= 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score, no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA) and no treatment failure. SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to Systemic Lupus Erythematosus (SLE), divided into 9 organ systems. For each organ system A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale =from 0(very well) to 100(very poor).
Time Frame: At Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 94 | 71 | 74 | 114
Participants | 50 | 44 | 48 | 77

12. Secondary Outcome: Cohort B: Number of Participants With Lupus Low Disease Activity State (LLDAS) Attainment at Week 24
Description: Lupus Low Disease Activity State (LLDAS) Attainment at Week 24 is defined as meeting all of the following criteria at the specified time point: SLE Disease Activity Index 2000 (SLEDAI-2K) ≤4 with no activity in major organ systems, no new disease activity compared to the previous assessment, Physician's Global Assessment (PGA) ≤1, current prednisone dose ≤7.5 mg/day, and standard maintenance dosing of immunosuppressive therapies. The number of participants with LLDAS Attainment at Week 24 were reported.
Time Frame: At Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 94 | 71 | 74 | 114
Participants | 23 | 21 | 32 | 35

13. Secondary Outcome: Cohort B: Number of Participants With Remission Attainment at Week 24
Description: Remission attainment was defined as a Clinical Hybrid Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus Disease Activity Index score of 0, Physician's Global Assessment of Systemic Lupus Erythematosus <0.5 (0-3 scale), daily prednisolone-equivalent dose ≤5 mg, and stable use of immunosuppressive therapies including biologics. Number of participants who attained remission was reported.
Time Frame: At Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 94 | 71 | 74 | 114
Participants | 10 | 7 | 8 | 20

14. Secondary Outcome: Cohort B: Percentage of Participants With 50% Reduction in Baseline Tender and Swollen Count at Week 24
Description: The 28-joint count questionnaire assesses 14 joints on each side (28 joints overall) for both tenderness and swelling. The outcome for the assessment of each joint can be "absent", "present", "replaced" or "unable to evaluate".Tender 28-joint count will be derived as the count of joints which are tender. Swollen 28-joint count will be derived as the count of joints which are swollen. The number of tender and swollen joints will be calculated as the count of joints which are both tender and swollen. Percentage of Participants with 50% Reduction in Baseline Tender and Swollen Count at Week 24 was reported.
Time Frame: At Week 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 65 | 46 | 54 | 79
percentage of participants | 68.8 | 72.2 | 77.6 | 79.1

15. Secondary Outcome: Cohort B: Time to First Moderate/Severe British Isles Lupus Assessment Group (BILAG) Flare
Description: Time to First Moderate/Severe British Isles Lupus Assessment Group (BILAG) Flare is defined as the time from baseline to the first occurrence of moderate or severe disease activity, as measured by the BILAG Index. The BILAG Index assesses clinical signs, symptoms, and laboratory parameters related to systemic lupus erythematosus (SLE) across 9 organ systems. Each organ system is scored alphabetically: A (severe disease), B (moderate disease), C (mild stable disease), D (inactive but previously active), and E (inactive and never affected). A moderate/severe flare is defined as the presence of at least one new or worsening BILAG A score (severe disease activity) or two or more new or worsening BILAG B scores (moderate disease activity) in any organ system, compared to the previous visit. Time to First Moderate/Severe British Isles Lupus Assessment Group (BILAG) Flare was estimated via Kaplan-Meier method.
Time Frame: Baseline (Day 1) through Week 24
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 94 | 71 | 74 | 114
days | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals. | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals. | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals. | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals.

16. Secondary Outcome: Cohort B: Time to First Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Flare Index (SFI) Severe Flare
Description: Time to First Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Flare Index (SFI) Severe Flare is defined as the time from baseline to the first occurrence of a severe flare, as measured by the SLEDAI Flare Index (SFI). A severe flare is characterized by a ≥12-point increase in the SLEDAI score from the previous visit, accompanied by a ≥2.5-point increase in the physician's global assessment (on a 0-3 visual analogue scale), and a change in treatment such as initiation of corticosteroids at a dose >0.5 mg/kg/day and/or the addition of a new immunosuppressive agent. Time to First Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Flare Index (SFI) Severe Flare was estimated via Kaplan-Meier method.
Time Frame: Baseline (Day 1) through Week 24
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 94 | 71 | 74 | 114
days | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals. | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals. | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals. | NA [NA to NA] — The number of events was insufficient to calculate the median and its associated 95% confidence intervals.

17. Secondary Outcome: Cohort A and B: Change From Baseline in Skindex 29+3 Symptom Domain Score at Week 24
Description: The Skindex 29+3 is a self-reported measure of skin-specific symptoms and functioning for CLE populations, and includes items from the Skindex-29, designed for use across dermatologic conditions, and 3 additional items specific for lupus. Subscale scores are generated for each of the 3 original domains of the Skindex-29 i.e., symptoms, functioning, and emotional well-being. For all subscale scores, higher scores indicate lower functioning/worse symptoms. The symptoms domain includes items measuring physical sensations such as itching, burning, stinging, and pain. Each item is rated on a 5-point Likert scale from 1 ("never") to 5 ("all the time"), and scores are transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Time Frame: Baseline and at week 24
Population: The FAS included all participants randomized in the cohort to which they were eligible."Overall number of participants analyzed" refers to those evaluable for the outcome measure. Participants who were randomized in error were excluded from FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 19 | 21 | 20 | 24 | 26 | 19 | 27 | 34
scores on a scale | -13.7 [-21.4 to -6.1] | -27.3 [-34.7 to -19.9] | -28.6 [-36.1 to -21.2] | -21.9 [-28.8 to -14.9] | -9.2 [-16.5 to -2.0] | -17.5 [-25.9 to -9.2] | -15.2 [-22.6 to -7.9] | -17.0 [-23.5 to -10.5]

18. Secondary Outcome: Cohort A and B: Change From Baseline in the Skindex 29+3 Functioning Domain Scores at Week 24
Description: The Skindex 29+3 is a self-reported measure of skin-specific symptoms and functioning for CLE populations, and includes items from the Skindex-29, designed for use across dermatologic conditions, and 3 additional items specific for lupus. Subscale scores are generated for each of the 3 original domains of the Skindex-29 i.e., symptoms, functioning, and emotional well-being. For all subscale scores, higher scores indicate lower functioning/worse symptoms. The functioning domain assesses the impact of skin disease on daily activities, social interactions, and work. Items are rated on a 5-point Likert scale (1 = "never" to 5 = "all the time") and transformed to a 0-100 scale, where higher scores reflect greater impairment in functioning.
Time Frame: Baseline and at Week 24
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 19 | 21 | 20 | 24 | 26 | 18 | 27 | 34
scores on a scale | -12.2 [-19.5 to -4.8] | -17.9 [-24.9 to -10.8] | -20.3 [-27.4 to -13.1] | -15.1 [-21.7 to -8.5] | -11.1 [-18.4 to -3.8] | -14.2 [-23.0 to -5.5] | -11.3 [-18.7 to -3.8] | -15.4 [-22.0 to -8.9]

19. Secondary Outcome: Cohort A and B: Change From Baseline in the Skindex 29+3 Emotion Domain Scores at Week 24
Description: The Skindex 29+3 is a self-reported measure of skin-specific symptoms and functioning for CLE populations, and includes items from the Skindex-29, designed for use across dermatologic conditions, and 3 additional items specific for lupus. Subscale scores are generated for each of the 3 original domains of the Skindex-29 i.e., symptoms, functioning, and emotional well-being. For all subscale scores, higher scores indicate lower functioning/worse symptoms. The emotion domain of the Skindex-29+3 assesses the psychological impact of skin disease in individuals with cutaneous lupus erythematosus. It includes items that measure feelings such as embarrassment, frustration, anger, sadness, and worry related to skin symptoms. Each item is rated on a 5-point Likert scale from 1 ("never") to 5 ("all the time"), and scores are transformed to a 0-100 scale, with higher scores indicating greater emotional distress.
Time Frame: Baseline and at Week 24
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 19 | 21 | 20 | 24 | 26 | 18 | 27 | 34
scores on a scale | -15.8 [-25.3 to -6.4] | -23.1 [-32.3 to -13.9] | -21.2 [-30.5 to -12.0] | -23.2 [-31.8 to -14.5] | -15.3 [-24.6 to -6.0] | -18.0 [-29.1 to -6.8] | -16.9 [-26.3 to -7.4] | -16.3 [-24.6 to -7.9]

20. Secondary Outcome: Cohort A and B: Change From Baseline in the Skindex 29+3 Lupus-Specific Domain Scores at Week 24
Description: The Skindex-29+3 is a self-reported measure of skin-specific symptoms and functioning for CLE populations. It includes items from the Skindex-29, designed for use across dermatologic conditions, and 3 additional items specific to lupus. Subscale scores are generated for the 3 original domains: symptoms, functioning, and emotional well-being. For all subscales, higher scores indicate worse symptoms or lower functioning. The lupus-specific domain captures symptoms and concerns unique to cutaneous lupus, including sensitivity to sunlight, flares from environmental exposure, and emotional impact of lupus-related skin changes. Each item is rated on a 5-point Likert scale from 1 ("never") to 5 ("all the time"), and scores are transformed to a 0-100 scale. Higher scores reflect greater symptom burden and disease impact.
Time Frame: Baseline and at Week 24
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 18 | 21 | 20 | 24 | 26 | 18 | 27 | 34
scores on a scale | -15.5 [-26.8 to -4.3] | -19.9 [-30.6 to -9.1] | -21.1 [-31.9 to -10.3] | -11.0 [-21.1 to -1.0] | -16.4 [-26.8 to -6.0] | -10.9 [-23.1 to 1.3] | -13.1 [-23.8 to -2.4] | -14.5 [-23.8 to -5.2]

21. Secondary Outcome: Cohort A and B: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scores at Week 24
Description: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) is a 13-item, self-reported questionnaire designed to assess fatigue and its impact on daily activities and functioning in individuals with chronic illness, including systemic lupus erythematosus. Each item is rated on a 5-point Likert-type scale ranging from 0 = "not at all" to 4 = "very much". Items are scored to ensure that 0 represents the worst and 4 the best possible outcome. The score ranges from 0 to 52, with higher scores indicating less fatigue and better functioning.
Time Frame: Baseline and at Week 24
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
Number analyzed (Participants) | 19 | 21 | 20 | 23 | 79 | 63 | 65 | 101
scores on a scale | 3.0 [0.3 to 5.8] | 2.0 [-0.7 to 4.7] | 6.9 [4.2 to 9.6] | 4.3 [1.7 to 6.8] | 2.4 [0.4 to 4.4] | 4.8 [2.5 to 7.0] | 3.6 [1.4 to 5.8] | 5.1 [3.3 to 6.9]

ADVERSE EVENTS:
Time Frame: From screening up to safety follow up period (up to approximately 33 weeks)
Description: Participants were included in the treatment group in which they actually received study treatment.
Arm/Group | Cohort A: Placebo | Cohort A: Enpatoran 25 mg | Cohort A: Enpatoran 50 mg | Cohort A: Enpatoran 100 mg | Cohort B (Part 1 + Part 2): Placebo | Cohort B (Part 2): Enpatoran 25 mg | Cohort B (Part 2): Enpatoran 50 mg | Cohort B (Part 1 + Part 2): Enpatoran 100 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/26 | 0/26 | 0/95 | 0/71 | 0/74 | 0/114
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/24 | 0/26 | 1/26 | 3/95 | 1/71 | 3/74 | 5/114
Other Adverse Events (participants affected / at risk) | 8/26 | 4/24 | 6/26 | 13/26 | 29/95 | 17/71 | 24/74 | 33/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Placebo (N=26) | Cohort A: Enpatoran 25 mg (N=24) | Cohort A: Enpatoran 50 mg (N=26) | Cohort A: Enpatoran 100 mg (N=26) | Cohort B (Part 1 + Part 2): Placebo (N=95) | Cohort B (Part 2): Enpatoran 25 mg (N=71) | Cohort B (Part 2): Enpatoran 50 mg (N=74) | Cohort B (Part 1 + Part 2): Enpatoran 100 mg (N=114)
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vein rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Placebo (N=26) | Cohort A: Enpatoran 25 mg (N=24) | Cohort A: Enpatoran 50 mg (N=26) | Cohort A: Enpatoran 100 mg (N=26) | Cohort B (Part 1 + Part 2): Placebo (N=95) | Cohort B (Part 2): Enpatoran 25 mg (N=71) | Cohort B (Part 2): Enpatoran 50 mg (N=74) | Cohort B (Part 1 + Part 2): Enpatoran 100 mg (N=114)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 7 | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4 | 5 | 6 | 7 | 9 | 8
Urinary tract infection (Infections and infestations) | 4 | 0 | 0 | 2 | 8 | 0 | 5 | 11
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 6 | 10
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 5 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT05162586/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT05162586/SAP_001.pdf